CLINICAL TRIAL: NCT01632891
Title: An Open-Label, Proof of Concept, Randomized Trial Comparing a LPV/r-Based to an nNRTI-Based Antiretroviral Therapy Regimen for Clearance of Plasmodium Falciparum Subclinical Parasitemia in HIV-infected Adults With CD4+ Counts >200 and <500 Cells/mm^3
Brief Title: Comparing PI-Based to a nNRTI-based ART for Clearance of Plasmodium Falciparum Parasitemia in HIV-Infected
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5297; 1U01AI068636 (NIH)
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: HIV-1 Infection; Pf Subclinical Parasitemia
MeSH Terms: interventions — Lopinavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; Nevirapine; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LPV/r-based ART (Experimental): Participants were prescribed to LPV/r-based antiretroviral therapy (ART) for 15 days, which includes lopinavir/ritonavir plus emtricitabine/tenofovir disoproxil fumarate; followed by an nNRTI-based ART, which includes efavirenz, nevirapine, plus emtricitabine/tenofovir disoproxil fumarate, and Trimethoprim/sulfamethoxazole prophylaxis to take from day 16 through day 30.
  Interventions: Drug: Lopinavir/ritonavir; Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Efavirenz; Drug: Nevirapine; Drug: Trimethoprim/sulfamethoxazole
- nNRTI-based ART (Experimental): Participants were prescribed to nNRTI-based ART for 15 days, which includes efavirenz, nevirapine, plus emtricitabine/tenofovir disoproxil fumarate, followed by an nNRTI-based ART and Trimethoprim/sulfamethoxazole prophylaxis to take from day 16 through day 30.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Efavirenz; Drug: Nevirapine; Drug: Trimethoprim/sulfamethoxazole

INTERVENTIONS:
Drug: Lopinavir/ritonavir — Participants received two 200 mg/50 mg tablets of lopinavir/ritonavir orally twice daily.
  Other Names: LPV/r
  Arms: LPV/r-based ART
Drug: Emtricitabine/tenofovir disoproxil fumarate — Participants received one 200 mg/300 mg tablet of Emtricitabine/tenofovir disoproxil fumarate orally once daily.
  Other Names: FTC/TDF
Drug: Efavirenz — Participants received one 600 mg tablet of efavirenz orally once daily.
  Other Names: EFV
Drug: Nevirapine — If unable to take efavirenz, participants received on 200 mg tablet of nevirapine orally once daily.
  Other Names: NVP
Drug: Trimethoprim/sulfamethoxazole — Participants received one 160 mg/800 mg tablet of trimethoprim/sulfamethoxazole orally once daily.
  Other Names: TMP/SMX

SUMMARY:
The purpose of this study was to see if antiretroviral therapy (ART) is safe and works at getting rid of malaria in blood and to see whether one type of ART is better than another. This study may offer information for further research in looking at whether ART plays a role in the prevention and treatment of malaria.

DETAILED DESCRIPTION:
A5297 was a Phase I/II, open-label, proof of concept, two-step, two-arm, randomized controlled clinical trial (RCT) to test the superiority of lopinavir/ritonavir (LPV/r)-based antiretroviral therapy (ART) to non-nucleoside reverse transcriptase (nNRTI)-based ART for clearance of Plasmodium falciparum (Pf) subclinical parasitemia (SCP).

The study consisted of two steps. At study Step 1 entry, participants were randomized 1:1 to either LPV/r-based ART or nNRTI-based ART for 15 days. In study Step 2, all participants received nNRTI-based ART and TMP/SMX prophylaxis for 15 days. The total study duration was 30 days.

Study visits occurred every 3 days in Step 1, and every 5 days in Step 2. At each study visit, 2 samples were taken for measurement of parasite density, except day 15 and day 30 at which 3 samples were taken.

Adverse events which occurred after randomization were also recorded. Signs/symptoms and diagnoses were evaluated at each visit, while safety labs (including Hemoglobin, hematocrit, white blood cell count (WBC), differential WBC, platelet count, and absolute neutrophil count (ANC), glucose, electrolytes (sodium, potassium, chloride, bicarbonate), total bilirubin, AST (SGOT), ALT (SGPT), albumin, alkaline phosphatase, and creatinine) were taken at day 15 and day 30, or if indicated at other study visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4+ count > 200 and < 500 cells/mm^3 obtained within 30 days prior to study entry at a DAIDS-approved laboratory.
* Pf SCP confirmed in a laboratory approved to conduct parasitemia microscopy. Note: Pf SCP defined as meeting all three of the following criteria within 72 hours prior to study entry:

  1. Microscopy confirmed parasitemia (see section 6.3.6 and the A5297 Manual of Procedures [MOPS])
  2. An oral temperature < 37.5°C.
  3. The absence of Grade 2 or greater signs or symptoms thought to be related to clinical malaria including:

     1. headache
     2. malaise or fatigue
     3. abdominal discomfort
     4. muscle or joint pain
     5. fever
     6. chills
     7. perspiration
     8. anorexia
     9. vomiting
     10. other signs or symptoms thought to be related to clinical malaria
* Certain laboratory values obtained within 14 days prior to study entry, as detailed in section 4.1.4 of the protocol.
* Hepatitis B surface antigen (HBsAg) negative within 30 days prior to entry.
* Female study volunteers of reproductive potential have a negative serum or urine pregnancy test performed within 72 hours prior to entry.
* All study volunteers agree not to participate in a conception process (eg, active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) for study duration. If participating in sexual activity that could lead to pregnancy, must agree to use two reliable forms of contraceptive simultaneously while receiving protocol-specified medications. One form of contraceptive must be a barrier method if a participant receives EFV. Participants must agree to continue the use of two contraceptives for 6 months after stopping EFV and 6 weeks after stopping all other protocol-specified medications.
* Study volunteers who are not of reproductive potential are eligible without requiring the use of a contraceptive.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* Willing and able to return to the clinic twice to three times a day for study visits.

Exclusion Criteria:

Step 1: Exclusion Criteria

* Previous history or current use of ART.
* Single dose NVP or dual therapies used for Prevention of mother-to-child transmission (PMTCT) within 2 years prior to entry.
* Use of any medication with antimalarial activity, including TMP/SMX (see list of prohibited medications in the A5297 Manual of Procedures (MOPS)), within 14 days prior to study entry.
* Confirmed or clinically suspected OIs (including but not limited to tuberculosis, clinical malaria, PCP), or other pulmonary or gastrointestinal infections for which potential participants did not complete treatment more than 30 days prior to enrollment or have signs and symptoms during screening.
* Breastfeeding.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.
* Results suggestive of active pulmonary disease from a chest x-ray performed within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2016-06-19 (Actual); Study Completion 2016-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnstone Kumwenda, FRCP, Study Chair — College of Medicine-Johns Hopkins Project; Douglas Shaffer, MD, MHS, Study Chair — Kenya Medical Research Institute/Walter Reed Project
Locations (5):
- Kenya (3):
  - AMPATH at Moi Univ. Teaching Hosp. Eldoret CRS (12601), Eldoret
  - Walter Reed Project - Kenya Med. Research Institute Kericho CRS (12501), Kericho
  - Kisumu Crs (31460), Kisumu
- College of Med. JHU CRS (30301), Blantyre, Malawi
- Joint Clinical Research Centre (JCRC) (12401), Kampala, Uganda

REFERENCES:
- [Derived] Shaffer D, Kumwenda J, Chen H, Akelo V, Angira F, Kosgei J, Tonui R, Ssali F, McKhann A, Hogg E, Stewart VA, Murphy SC, Coombs R, Schooley R; A5297 Team. Brief Report: No Differences Between Lopinavir/Ritonavir and Nonnucleoside Reverse Transcriptase Inhibitor-Based Antiretroviral Therapy on Clearance of Plasmodium falciparum Subclinical Parasitemia in Adults Living With HIV Starting Treatment (A5297). J Acquir Immune Defic Syndr. 2022 Feb 1;89(2):178-182. doi: 10.1097/QAI.0000000000002839. PMID 34693933
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 — http://rsc.tech-res.com/safetyandpharmacovigilance/
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/safetyandpharmacovigilance/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 clinics in Africa. The first participant enrolled on January 10, 2014. The last participant enrolled on May 20, 2016.
Period: Overall Study
Arm/Group | LPV/R-based ART | nNRTI-based ART
Started | 26 | 26
Completed | 25 | 25
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | LPV/R-based ART | nNRTI-based ART | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [24 to 38] | 31 [24 to 39] | 31 [24 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 17 | 18 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 26 | 26 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 1 | 1 | 2
  Uganda | 1 | 0 | 1
  Kenya | 24 | 25 | 49
CD4 cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 360 [265 to 407] | 302 [256 to 389] | 324 [259 to 404]
Log10(HIV-1 RNA) [Median (Inter-Quartile Range); unit: Log10(cp/ml)] | 5.11 [4.65 to 5.51] | 5.37 [4.56 to 5.76] | 5.18 [4.60 to 5.71]
Log10(parasite density) [Median (Inter-Quartile Range); unit: Log10(parasites/µL)] | 2.69 [2.08 to 3.40] | 2.50 [1.66 to 3.26] | 2.66 [1.92 to 3.35]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Plasmodium Falciparum (Pf) Subclinical Parasitemia (SCP) Clearance
Description: Pf SCP clearance defined by polymerase chain reaction (PCR) < 10 parasites/µL on three consecutive occasions within a 24-hour period.
  If a participant had missing data on day 15, they were considered as not having clearance.
Time Frame: Day 15 (3 samples collected, separated by at least 5 hours and all three collected within 24-hours)
Population: Primary analysis is based on intent-to-treat principles and includes all randomized participants.
Measure: Number; unit: Proportion of participants
Arm/Group | LPV/R-based ART | nNRTI-based ART
Number analyzed (Participants) | 26 | 26
Proportion of participants
  Proportion Cleared | 0.23 | 0.27
  Proportion Not Cleared | 0.77 | 0.73
Statistical Analysis 1: Comparison: LPV/R-based ART vs nNRTI-based ART; Compare proportions of Pf SCP clearance between treatment arms; Test type: Superiority — Test used alpha level of 0.05; p = 1.00, Fisher Exact

2. Secondary Outcome: Time to First Pf SCP Clearance
Description: Time to clearance is defined by time to first measurement with PCR < 10 parasites/µL, and is evaluated as the point estimate and 95% CI for the day when 50% of participants cleared parasite.
Time Frame: From study entry up to day 30
Population: Analysis only includes participants who received 15 days of treatment, excluding one participant on LPV/r-based ART.
  One participant on nNRTI-based ART had missing data at all time points.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | LPV/R-based ART | nNRTI-based ART
Number analyzed (Participants) | 25 | 25
Days | 12 [5 to 29] | 14 [2 to 29]

3. Secondary Outcome: Log10(Pf Parasite Density)
Description: Pf parasite density was determined by PCR. If parasite density equals 0, the value is set to 0.01 before log10 transformation. The value 0.01 was chosen based on the smallest observed parasite density value of 0.017.
Time Frame: Entry, days 3, 6, 9, 12, 15, 20, 25, 30
Population: Analysis only includes participants who received 15 days of treatment, excluding one participant on LPV/r-based ART.
  One participant on nNRTI-based ART had missing data at all time points. Several samples were missing at various time points, as shown by number of participants for each day.
Measure: Mean (95% Confidence Interval); unit: log10(parasites/µL)
Arm/Group | LPV/R-based ART | nNRTI-based ART
Number analyzed (Participants) | 25 | 25
log10(parasites/µL)
  Entry: number analyzed (Participants) | 25 | 24
  Entry | 2.48 [1.93 to 3.02] | 2.09 [1.32 to 2.85]
  Day 3: number analyzed (Participants) | 25 | 24
  Day 3 | 1.92 [1.40 to 2.44] | 1.57 [0.77 to 2.37]
  Day 6: number analyzed (Participants) | 24 | 23
  Day 6 | 1.77 [1.24 to 2.29] | 1.49 [0.65 to 2.33]
  Day 9: number analyzed (Participants) | 24 | 21
  Day 9 | 1.65 [1.03 to 2.27] | 1.63 [0.85 to 2.41]
  Day 12: number analyzed (Participants) | 23 | 23
  Day 12 | 1.59 [0.99 to 2.19] | 1.56 [0.66 to 2.46]
  Day 15: number analyzed (Participants) | 25 | 23
  Day 15 | 1.59 [1.00 to 2.18] | 1.43 [0.63 to 2.23]
  Day 20: number analyzed (Participants) | 24 | 20
  Day 20 | 0.65 [0.05 to 1.25] | 0.67 [-0.19 to 1.52]
  Day 25: number analyzed (Participants) | 24 | 22
  Day 25 | 0.28 [-0.42 to 0.99] | 0.49 [-0.36 to 1.33]
  Day 30: number analyzed (Participants) | 25 | 23
  Day 30 | 0.14 [-0.51 to 0.79] | 0.30 [-0.35 to 0.95]

4. Secondary Outcome: Change in log10(Pf Parasite Density) From Entry to Day 30
Description: Change is evaluated as log10(Pf parasite density) at day 30 minus log10(Pf parasite density) at entry.
  Change is evaluated in four groups:
  * Randomized to nNRTI-based ART with continued Pf SCP at day 15
  * Randomized to nNRTI-based ART with clearance of Pf SCP at day 15
  * Randomized to LPV/r-based ART with continued Pf SCP at day 15
  * Randomized to LPV/r-based ART with clearance of Pf SCP at day 15
Time Frame: Entry, Day 30
Population: All participants enrolled with results available at entry and day 30:
  3 participants were missing data in 'nNRTI-based ART, not cleared' group.
  1 participant was missing data in 'nNRTI-based ART, cleared' group.
  1 participant was missing data in 'LPV/r-based ART, not cleared' group.
Measure: Median (Inter-Quartile Range); unit: log10(parasites/µL)
Groups:
- nNRTI-based ART, Not Cleared: Randomized to nNRTI based ART with continued Pf SCP at day 15
- nNRTI-based ART, Cleared: Randomized to nNRTI based ART with clearance of Pf SCP at day 15
- LPV/R-based ART, Not Cleared: Randomized to LPV/r based ART with continued Pf SCP at day 15
- LPV/R-based ART, Cleared: Randomized to LPV/r based ART with clearance of Pf SCP at day 15
Arm/Group | nNRTI-based ART, Not Cleared | nNRTI-based ART, Cleared | LPV/R-based ART, Not Cleared | LPV/R-based ART, Cleared
Number analyzed (Participants) | 16 | 6 | 19 | 6
log10(parasites/µL) | -2.26 [-3.30 to -1.29] | -1.65 [-3.39 to 0.40] | -1.82 [-3.65 to -0.39] | -3.61 [-4.96 to -2.19]

5. Secondary Outcome: Number of Participants With Uncomplicated Clinical Malaria
Description: Uncomplicated clinical malaria is defined as the presence of non-severe fever/symptoms and parasitemia without organ complication.
Time Frame: From study entry to day 30
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | LPV/R-based ART | nNRTI-based ART
Number analyzed (Participants) | 26 | 26
Participants | 2 | 1

6. Secondary Outcome: Number of Participants With Detectable Pf Gametocyte Density
Description: Number of participants with detectable Pf gametocyte density as determined by PCR. Due to the large number of undetectable results, this outcome was measured as dichotomous.
Time Frame: Entry, days 3, 6, 9, 12, 15, 20, 25, 30
Population: Analysis only includes participants who received 15 days of treatment, excluding one participant on LPV/r-based ART.
  One other participant on LPV/r-based ART had missing data at all time points. Several samples were missing at various time points, as shown by number of participants for each day.
Measure: Count of Participants; unit: Participants
Arm/Group | LPV/R-based ART | nNRTI-based ART
Number analyzed (Participants) | 24 | 26
Participants
  Entry: number analyzed (Participants) | 23 | 25
  Entry | 11 | 12
  Day 3: number analyzed (Participants) | 24 | 25
  Day 3 | 10 | 15
  Day 6: number analyzed (Participants) | 23 | 24
  Day 6 | 9 | 12
  Day 9: number analyzed (Participants) | 24 | 22
  Day 9 | 11 | 13
  Day 12: number analyzed (Participants) | 23 | 25
  Day 12 | 6 | 11
  Day 15 | 10 | 14
  Day 20: number analyzed (Participants) | 23 | 24
  Day 20 | 11 | 14
  Day 25: number analyzed (Participants) | 24 | 25
  Day 25 | 12 | 16
  Day 30: number analyzed (Participants) | 24 | 24
  Day 30 | 11 | 13

7. Secondary Outcome: Change in log10(Pf Gametocyte Density) From Entry to Day 30
Description: Change in log10(Pf gametocyte density) as evaluated using a Hodges-Lehmann estimate from entry to day 30 is evaluated in two groups:
  * Randomized to nNRTI-based ART with continued Pf SCP at day 15
  * Randomized to LPV/r-based ART with continued Pf SCP at day 15
  Analysis was not conducted in either group with clearance at day 15 due to the small sample size and high number of undetectable samples in both clearance groups at entry and day 30.
Time Frame: Entry, Day 30
Population: All participants with results available at both entry and day 30 who did not have Pf SCP clearance at day 15.
  1. participant was missing from the nNRTI-based ART, not cleared group
  2. participants were missing from the LPV/r-based ART, not cleared group
Measure: Number (95% Confidence Interval); unit: log10(gametocyte/µL)
Arm/Group | nNRTI-based ART, Not Cleared | nNRTI-based ART, Cleared | LPV/R-based ART, Not Cleared | LPV/R-based ART, Cleared
Number analyzed (Participants) | 18 | 0 | 18 | 0
log10(gametocyte/µL) | -0.46 [-1.33 to 0.20] |  | 0.17 [-0.75 to 0.89] |

ADVERSE EVENTS:
Time Frame: From randomization to study completion at 30 days
Description: The following adverse event information was collected:
  * Signs and symptoms Grade ≥ 3, and signs and symptoms that led to a change in treatment regardless of grade
  * All laboratory values Grade ≥ 2, and laboratory values that led to a change in treatment regardless of grade
  * All diagnoses identified by ACTG criteria for clinical events and other diseases
  * Deaths Grading performed according to DAIDS AE Grading Table (V1.0). SAEs defined in EAE Manual (V2.0). Refer to Protocol Section 11.
Arm/Group | LPV/R-based ART | nNRTI-based ART
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 3/26 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/R-based ART (N=26) | nNRTI-based ART (N=26)
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 1
Plasmodium falciparum infection (Infections and infestations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights